CLINICAL TRIAL: NCT06534112
Title: Evaluation of Short-term Changes and Self-reported User Experiences Related to the Know Your OQ™ Initiative
Brief Title: Evaluation of the Know Your OQ™ Oral Health Literacy Tool in an Indian Population
Acronym: KYOQIN
Status: Completed | Type: Observational
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Other Study IDs: CRO-2024-03-KYOQ-BG
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-07

CONDITIONS: Oral Health Literacy
Keywords: Oral Health Quotient; KYOQ; Oral Health Education

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Regular Consumers
- Nurses

SUMMARY:
This was a research study to evaluate the effectiveness of the questionnaire "Know Your OQ™" (Know Your Oral Health Quotient™) in changing people's level of knowledge about oral health in India and to evaluate the readability, understanding and ease of completion of the questionnaire "Know Your OQ™".

ELIGIBILITY:
Inclusion Criteria:

* Sign Informed Consent Form
* Male and female subjects aged ≥18 years old
* Availability of 10 days for completing the study
* Belong to NCCS (National Consumer Classification System) A,B
* Access to a cell phone, laptop, tablet or computer with internet/data connection
* Fluent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 150 male and female adults were split into two groups: 100 regular subjects and 50 nurses. These groups were further stratified by educational qualification (Completed High School, Pursuing Graduation, Completed Graduation, Completed Post Graduation), sex (male and female), age group (18-24, 25-35, 36-45, 46-55, 56-65, >65), experience with oral health problems (yes and no), and the cities they reside in (Mumbai, Delhi, Chennai, Kolkata, Bengaluru).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-06-08 (Actual); Study Completion 2024-06-08 (Actual)

PRIMARY OUTCOMES:
Changes in Knowledge, Attitude, Practice (KAP) | Baseline, Intervention, Immediate Follow-Up, 1 week Follow-Up
  Change in Knowledge, Attitude, and Practice before and after exposure to the Know Your OQ™ tool. Day minus 3: Pretest Knowledge, Attitude, Practice (KAP) & Demographics, Day 0: Know Your OQ, Day 0 Immediate follow up: Post-test Comprehension Questionnaire, Week 1 follow up: Post test Knowledge, Attitudes and Practices Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- IPSOS Research Private Limited, Mumbai, India